CLINICAL TRIAL: NCT04657536
Title: Randomized Multicenter Clinical Trial for Evaluating the Efficacy of Temperature-controlled Radiofrequency Compared With Topical Estriol in the Treatment of Vulvovaginal Atrophy in Postmenopausal Women
Brief Title: Evaluating the Efficacy of Temperature-controlled Radiofrequency (TRF) in the Treatment of Vulvovaginal Atrophy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Chinese Association of Plastics and Aesthetics (Unknown)
Responsible Party: Principal Investigator, Zhaolijun, associate professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 2.0；20200221
Record Dates: First submitted 2020-10-08; First posted 2020-12-08 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Postmenopausal Vulvovaginal Atrophy
Keywords: vulvovaginal atrophy; temperature-controlled radiofrequency; postmenopausal woman; Genitourinary Syndrome of Menopause
MeSH Terms: interventions — Estriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRF group (Experimental): the group who treated with temperature controlled radiofrequency
  Interventions: Device: high frequency fulguration equipment
- Estriol group (Active Comparator): the group who treated with promestriene vaginal soft capsules
  Interventions: Drug: promestriene vaginal soft capsules

INTERVENTIONS:
Device: high frequency fulguration equipment — All subjects will be carried out with 3 standard protocol TRF treatments to the vulvovaginal tissue using the high frequency fulguration equipment (Shenzhen Peninsula Medical co., Ltd) at 10-day to 15-day intervals. Radiofrequency energy was applied to the vaginal canal through a specialized probe combining monopolar and bipolar treatment modes. Monopolar treatment mode is for 15 minutes. Aim the three indication points A, B and C on the probe to the direction of 12 o'clock in turn. Each area should be treated for about 5 minutes. Rotate the probe clockwise when changing the area for treatment.Bipolar treatment mode is for 10 minutes. Firstly, indication point A is aimed to 12 o'clock for 5-minutes treatment and then the probe is rotated 90°clockwise for another 5-minutes treatment. The power setting will be 35-40w, and the target temperature setting will be 40 to 45℃, titrated to subject tolerance.
  Other Names: temperature controlled radiofrequency
  Arms: TRF group
Drug: promestriene vaginal soft capsules — Promestriene vaginal soft capsules（Zhejiang Anbao Pharmaceutical Co. LTD）will be used 10mg once a day for continuous 20 days.
  Other Names: Estriol
  Arms: Estriol group

SUMMARY:
This project will be a prospective, multicenter, randomized cohort study. The investigators will select patients with vulvovaginal atrophy who have indications for treatment, and set up the experimental group (Peninsula temperature-controlled radiofrequency therapeutic apparatus group) and the control group (promestriene vaginal soft capsules group). Changes in vaginal exfoliated cell maturity index (MV), score of vaginal symptoms and signs, vaginal health index score (VHIS), female sexual function index score (FSFI), visual analogue score (VAS) before and after treatment, and adverse effects will be observed to analyze the safety and efficacy of temperature-controlled radiofrequency therapy for vulvovaginal atrophy in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal time at least one year.
* Genitourinary Syndrome of Menopause (GSM) related symptoms with moderate or severe intensity, such as dryness and dyspareunia, etc.
* Blood FSH≥30 IU/L (30mIU/mL)。
* Clinical symptoms and signs of vaginal atrophy score≥15.
* Breast ultrasound examination was grade 1-3 within 9 months before the study.
* Voluntary participation in clinical trials and signed informed consent.
* Patients followed the treatment regimen and completed the study.

Exclusion Criteria (one of the following criteria is excluded) :

* The patients who did not meet the inclusion criteria
* Received Estrogen replacement therapy (including local and systemic medication) within 3 months.
* Received any medicine (such as Baofukang suppository) to treat vulvovaginal atrophy within 3 months.
* Corticosteroids were used within 6 weeks. Long-term corticosteroids were used (intermittent nasal or skin application, eye drops and ears are allowed).
* Other experimental drugs were used within 1 month.
* Received vaginal laser therapy within 6 months.
* Patients with acute urinary tract infection;
* Patients with acute genital tract infection (genital herpes, trichomonad, fungal vaginitis; gonococcus, mycoplasma, chlamydia infection and bacterial vaginosis, etc.);
* Patients with pelvic organ prolapse greater than or equal to stage II;
* Patients with metal intrauterine device (IUD)；
* Patients with precancerous lesions or malignant tumors of vagina and cervix;
* Patients with serious heart, liver, brain, kidney, endocrine diseases, etc.
* Allergic to control drug and excipients.
* Other malignancies are known or suspected.
* With estrogen-dependent neoplasm.
* Confirm a history of depression or serious mental illness.
* There were consciousness barriers and communication barriers that could not cooperate with the experiment.
* Patients considered unsuitable for this clinical trial.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The change value of vaginal maturation index (VMI) compared with baseline | The two groups will be visited on day 0, 1 month and 3 months after the last treatment.
  The Vaginal Maturation Index (VMI) is an assessment done to establish the oestrogen effect in the body. The vaginal cytology specimens were collected from the mid-vaginal-wall before treatment and fixed in ThinPrep solution. The VMI is a ratio obtained with three main cell types found in the vaginal walls: parabasal cells(P), Intermediate cells (I) and superficial cells(S). The findings will be presented in a 0/0/0 format. VMI = [1 × (% superficial cells)] + [0.6 × (% intermediate cells)] + [0.2 × (% parabasal cells)]. This index enabled us to objectively evaluate the differential count of each cell group expressed as a percentage. The greater the degree of vaginal atrophy, the greater the estrogen deficiency. When at most 30% of the deep cells were present in the vaginal smears, mild hypoestrogenism was diagnosed. A deep cell percentage between 30% and 49% indicated moderate hypoestrogenism and a more than 50% deep cell percentage indicated hypoestrogenism.
the changes of vaginal symptoms and signs scores compared with baseline | The two groups will be visited on day 0, day 20（the control group is day 21），1 month and 3 months after the last treatment.
  Symptoms (vaginal dryness, pruritus, burning, pain, shallow dyspareunia, deep dyspareunia) will be individually scored by women and signs (vaginal mucosa and petechia, vaginal elasticity, mucosal luster) will be individually scored by the investigators as 0 = absence, 1 = mild, 2 = moderate, and 3 = severe alteration. In addition, a composite score of symptoms and signs will calculated by the addition of the intensity scores of all individual symptoms and signs (range, 0-27: The higher the score is, the more severe the genitourinary atrophy is.). Symptoms and signs score (SSC) will be obtained at each visiting to assess the effect of treatment on all individual.

SECONDARY OUTCOMES:
The changes of vaginal health index score (VHI) compared with baseline | The two groups will be visited on day 0, day 20（the control group is day 21），1 month and 3 months after the last treatment.
  VHI scores accounted for the following five parameters: elasticity, fluid volume, pH, epithelial integrity, and moisture. Each parameter will be graded from 1 (worst condition) to 5 (best condition) with a maximum possible score of 25 points. Scores less than 15 are indicative of vaginal atrophy.
The changes of female sexual function index score (FSFI) compared with baseline | The two groups will be visited on day 0, 1 month and 3 months after the last treatment.
  Sexual function will be measured using the Female Sexual Function Index (FSFI). This questionnaire, which contains 19 items, was developed as a brief, but multidimensional, self-reporting instrument to assess the key dimensions of female sexual function. It was developed based on a group of normal female controls and age-matched women who met the DSM-IV-TR criteria for female sexual arousal disorder (FSAD). The FSFI addresses six domains of sexual function (desire, arousal, lubrication, orgasm, satisfaction, and pain) and provides full-scale scores ranging from 2.0 (severe dysfunction) to 36.0 (absence of dysfunction). The validated FSFI version for the Chinese language will be used. A cutoff score of 26.55 will be used to differentiate the presence or absence of sexual dysfunction.
The changes of visual analogue score (VAS) compared with baseline | The two groups will be visited on day 0, day 20（the control group is day 21），1 month and 3 months after the last treatment.
  The Visual Analogue Scale (VAS) is a popular tool for the measurement of pain. The pain is represented by 11 Numbers from 0 to 10, 0 is painless and 10 is the most painful. The patient chooses one of these 11 Numbers to represent the pain level according to her own pain level.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No